CLINICAL TRIAL: NCT01082406
Title: A Single Centre, Randomised, Double-blind, Cross-over Trial in Healthy Male Subjects Investigating Bioequivalence and Pharmacokinetics of rFXIII (Avecia DS) to rFXIII (Novo Nordisk DS)
Brief Title: Comparison of a Blood Clotting Drug (Recombinant Factor XIII) Produced by Two Different Manufacturers in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1841-3788; 2009-016438-28 (EudraCT Number); U1111-1113-2008 (Other: WHO)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency; Healthy
MeSH Terms: interventions — recombinant factor XIII-A2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Experimental)
  Interventions: Drug: catridecacog
- Trial part 2 (Experimental)
  Interventions: Drug: recombinant factor XIII

INTERVENTIONS:
Drug: catridecacog — Single dose of 35 IU/kg body weight recombinant factor XIII (catridecacog) (Novo Nordisk) administered iv (into the vein) followed by a single dose of 35 IU/kg body weight recombinant factor XIII (Avecia) administered iv.
  Arms: Trial part 1
Drug: recombinant factor XIII — Single dose of 35 IU/kg body weight recombinant factor XIII (Avecia) to be administered iv (into the vein) followed by a single dose of 35 IU/kg body weight recombinant factor XIII (catridecacog) (Novo Nordisk) administered iv.
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to compare the metabolism of a blood-clotting drug (recombinant Factor XIII)) produced by two different manufacturers (Novo Nordisk and Avecia) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 30 kg/m2
* Good general health based on assessment of medical history, physical examination, ECG (electrocardiogram), and clinical laboratory data at screening, as judged by the physician
* Non-smokers

Exclusion Criteria:

* Known history of thromboembolic event(s) or potential thromboembolic risk as judged by the physician
* Blood transfusion within 3 months of trial start
* Positive for hepatitis B or C infection
* Positive for Human Immunodeficiency Virus (HIV) infection
* Excessive consumption of a diet deviating from a normal diet as judged by the physician
* Blood or plasma donation within the last 3 months prior to trial start
* Subjects with any history of migraine

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Plasma concentration-time curve (Area under Curve 0-28 days) for factor XIII activityfor both drug substances measured by the Berichrom® assay | after 4 weeks of treatment

SECONDARY OUTCOMES:
Number of adverse events (serious and non-serious) | over 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Harrow, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com